CLINICAL TRIAL: NCT02128932
Title: Efficacy and Safety of Semaglutide Once Weekly Versus Insulin Glargine Once Daily as Add on to Metformin With or Without Sulphonylurea in Insulin-naïve Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Semaglutide Once Weekly Versus Insulin Glargine Once Daily as add-on to Metformin With or Without Sulphonylurea in Insulin-naïve Subjects With Type 2 Diabetes
Acronym: SUSTAIN™ 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-3625; 2013-004392-12 (EudraCT Number); U1111-1146-0211 (Other: WHO); NL47781.018.14 (Registry Identifier: National Registry in The Netherlands)
Record Dates: First submitted 2014-04-24; First posted 2014-05-01 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Semaglutide 0.5 mg/week (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 1.0 mg/week (Experimental)
  Interventions: Drug: semaglutide
- Insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: semaglutide — Injected subcutaneously (under the skin) once weekly. Following 4 doses (4 weeks) of 0.25 mg semaglutide weekly subjects will receive 0.5 mg semaglutide weekly for 26 weeks.
  Arms: Semaglutide 0.5 mg/week; Semaglutide 1.0 mg/week
Drug: insulin glargine — Injected subcutaneously (under the skin) once daily. Subjects will start on 10 IU once daily and the dose will be adjusted according to fasting plasma glucose.
  Arms: Insulin glargine

SUMMARY:
This trial is conducted in Africa, North and South America, Asia and Europe. The purpose of the trial is to compare the effect of once-weekly dosing of two dose levels of semaglutide versus insulin glargine once-daily on glycaemic control after 30 weeks of treatment in insulin-naïve subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older at the time of signing informed consent
* Insulin-naïve subjects diagnosed with type 2 diabetes and on stable diabetes treatment with metformin or metformin and SU (metformin 1500 mg or higher or maximum tolerated dose and SU half of maximum allowed dose according to national label or higher) for at least 90 days before screening. Stable is defined as unchanged medication and unchanged dose
* HbA1c 7.0 - 10.0% (53 - 86 mmol/mol) both inclusive

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or of childbearing potential not using adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice) throughout the trial including the 5 week follow-up period
* Any disorder which, in the opinion of the Investigator might jeopardise subject's safety or compliance with the protocol
* Treatment with any glucose lowering agent(s) other than stated in the inclusion criteria in a period of 90 days before screening. An exception is short-term treatment (7 days or less in total) with insulin in connection with intercurrent illness
* History of chronic or idiopathic acute pancreatitis
* Screening calcitonin value greater than or equal to 50 ng/L
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome 2
* Severe renal impairment defined as estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73 m^2 per modification of diet in renal disease (MDRD) formula (4 variable version)
* Acute coronary or cerebrovascular event within 90 days before randomisation
* Heart failure, New York Heart Association Class IV
* Known proliferative retinopathy or maculopathy requiring acute treatment according to the opinion of the investigator
* Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer)
* Mental inability, unwillingness or language barrier precluding adequate understanding of or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2015-09-03 (Actual); Study Completion 2015-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (209):
- United States (120):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Ozark, Alabama
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Gilbert, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Carmichael, California
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Elk Grove, California
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Oceanside, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Pomona, California
  - Novo Nordisk Investigational Site, Rialto, California
  - Novo Nordisk Investigational Site, Rolling Hills Estates, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Sherman Oaks, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Lakeland, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, Spring Hill, Florida
  - Novo Nordisk Investigational Site, Winter Haven, Florida
  - Novo Nordisk Investigational Site, Winter Park, Florida
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Johns Creek, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Norcross, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Park City, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Lake Charles, Louisiana
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Natchitoches, Louisiana
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Sterling Heights, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Trenton, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Morganton, North Carolina
  - Novo Nordisk Investigational Site, Shelby, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Canal Fulton, Ohio
  - Novo Nordisk Investigational Site, Carlisle, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Corvallis, Oregon
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Clairton, Pennsylvania
  - Novo Nordisk Investigational Site, Jersey Shore, Pennsylvania
  - Novo Nordisk Investigational Site, Lansdale, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Gaffney, South Carolina
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Rapid City, South Dakota
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Humble, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, Marshall, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Wenatchee, Washington
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Godoy Cruz
- Croatia (4):
  - Novo Nordisk Investigational Site, Čakovec
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Krapinske Toplice
  - Novo Nordisk Investigational Site, Zagreb
- France (19):
  - Novo Nordisk Investigational Site, Bobigny
  - Novo Nordisk Investigational Site, Bois-Guillaume
  - Novo Nordisk Investigational Site, Bourgoin
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Marseille Cédex 05
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Pierre-Bénite
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Rang-du-Fliers
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Saint-Nazaire
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Trinité - La Martinique
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (12):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Jerichow
  - Novo Nordisk Investigational Site, Lampertheim
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Rostock
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Wangen
- India (10):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mysore, Karnataka
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Kolkata
  - Novo Nordisk Investigational Site, New Delhi
- Mexico (4):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Distrito Federal, México, D.F.
  - Novo Nordisk Investigational Site, México D.F., México, D.F.
  - Novo Nordisk Investigational Site, Aguascalientes
- Netherlands (3):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Hoofddorp
  - Novo Nordisk Investigational Site, Rotterdam
- North Macedonia (2):
  - Novo Nordisk Investigational Site, Skopje
  - Novo Nordisk Investigational Site, Tetovo
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Romania (5):
  - Novo Nordisk Investigational Site, Piteşti, Argeş
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Iași
- Slovakia (5):
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
  - Novo Nordisk Investigational Site, Piešťany
  - Novo Nordisk Investigational Site, Púchov
  - Novo Nordisk Investigational Site, Trenčín
- Slovenia (3):
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Ljubljana
  - Novo Nordisk Investigational Site, Novo Mesto
- South Africa (4):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- United Kingdom (13):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Harrogate, North Yorkshire
  - Novo Nordisk Investigational Site, Haxey
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Ipswich
  - Novo Nordisk Investigational Site, Northwood
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Sidcup
  - Novo Nordisk Investigational Site, Soham
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Taunton

REFERENCES:
- [Background] Rodbard HW, Bellary S, Hramiak I, Seino Y, Silver R, Damgaard LH, Nayak G, Zacho J, Aroda VR. GREATER COMBINED REDUCTIONS IN HbA1C >/=1.0% AND WEIGHT >/=5.0% WITH SEMAGLUTIDE VERSUS COMPARATORS IN TYPE 2 DIABETES. Endocr Pract. 2019 Jun;25(6):589-597. doi: 10.4158/EP-2018-0444. Epub 2019 Mar 13. PMID 30865526
- [Result] Aroda VR, Bain SC, Cariou B, Piletic M, Rose L, Axelsen M, Rowe E, DeVries JH. Efficacy and safety of once-weekly semaglutide versus once-daily insulin glargine as add-on to metformin (with or without sulfonylureas) in insulin-naive patients with type 2 diabetes (SUSTAIN 4): a randomised, open-label, parallel-group, multicentre, multinational, phase 3a trial. Lancet Diabetes Endocrinol. 2017 May;5(5):355-366. doi: 10.1016/S2213-8587(17)30085-2. Epub 2017 Mar 23. PMID 28344112
- [Result] Kapitza C, Dahl K, Jacobsen JB, Axelsen MB, Flint A. Effects of semaglutide on beta cell function and glycaemic control in participants with type 2 diabetes: a randomised, double-blind, placebo-controlled trial. Diabetologia. 2017 Aug;60(8):1390-1399. doi: 10.1007/s00125-017-4289-0. Epub 2017 May 19. PMID 28526920
- [Result] Warren M, Chaykin L, Trachtenbarg D, Nayak G, Wijayasinghe N, Cariou B. Semaglutide as a therapeutic option for elderly patients with type 2 diabetes: Pooled analysis of the SUSTAIN 1-5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2291-2297. doi: 10.1111/dom.13331. Epub 2018 Jun 7. PMID 29687620
- [Result] Ahren B, Atkin SL, Charpentier G, Warren ML, Wilding JPH, Birch S, Holst AG, Leiter LA. Semaglutide induces weight loss in subjects with type 2 diabetes regardless of baseline BMI or gastrointestinal adverse events in the SUSTAIN 1 to 5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2210-2219. doi: 10.1111/dom.13353. Epub 2018 Jun 12. PMID 29766634
- [Result] DeVries JH, Desouza C, Bellary S, Unger J, Hansen OKH, Zacho J, Woo V. Achieving glycaemic control without weight gain, hypoglycaemia, or gastrointestinal adverse events in type 2 diabetes in the SUSTAIN clinical trial programme. Diabetes Obes Metab. 2018 Oct;20(10):2426-2434. doi: 10.1111/dom.13396. Epub 2018 Jul 9. PMID 29862621
- [Result] Aroda VR, Ahmann A, Cariou B, Chow F, Davies MJ, Jodar E, Mehta R, Woo V, Lingvay I. Comparative efficacy, safety, and cardiovascular outcomes with once-weekly subcutaneous semaglutide in the treatment of type 2 diabetes: Insights from the SUSTAIN 1-7 trials. Diabetes Metab. 2019 Oct;45(5):409-418. doi: 10.1016/j.diabet.2018.12.001. Epub 2019 Jan 4. PMID 30615985
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Capehorn M, Ghani Y, Hindsberger C, Johansen P, Jodar E. Once-Weekly Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Common OAD: a Subgroup Analysis from SUSTAIN 2-4 and 10. Diabetes Ther. 2020 May;11(5):1061-1075. doi: 10.1007/s13300-020-00796-z. Epub 2020 Mar 19. PMID 32193837
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- [Derived] DeSouza C, Cariou B, Garg S, Lausvig N, Navarria A, Fonseca V. Efficacy and Safety of Semaglutide for Type 2 Diabetes by Race and Ethnicity: A Post Hoc Analysis of the SUSTAIN Trials. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz072. doi: 10.1210/clinem/dgz072. PMID 31769496
- [Derived] Jendle J, Birkenfeld AL, Polonsky WH, Silver R, Uusinarkaus K, Hansen T, Hakan-Bloch J, Tadayon S, Davies MJ. Improved treatment satisfaction in patients with type 2 diabetes treated with once-weekly semaglutide in the SUSTAIN trials. Diabetes Obes Metab. 2019 Oct;21(10):2315-2326. doi: 10.1111/dom.13816. Epub 2019 Jul 12. PMID 31215727
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at196 sites in 14 countries. Argentina: 3 sites; Croatia: 3 sites; France: 5 sites; Germany: 11 sites; India: 12 sites; Macedonia: 3 sites; Mexico: 3 sites; Netherlands: 3 sites; Romania: 5 sites; Slovakia: 5 sites; Slovenia:3 sites; South Africa: 4 sites; United Kingdom: 13 sites; United States: 123 sites.
Pre-assignment Details: Insulin-naïve subjects diagnosed with type 2 diabetes and on stable diabetes treatment with metformin or metformin and SU (metformin ≥1500 mg or maximum tolerated dose and SU≥ half of maximum allowed dose according to national label) for at least 90 days before screening. Stable is defined as unchanged medication and unchanged dose.
Groups:
- Semaglutide 0.5mg/Week: Subjects on semaglutide followed a fixed dose-escalation. The maintenance dose of 0.5 mg was to be reached after 4 doses (4 weeks) of 0.25 mg semaglutide. Doses could not be changed during the trial after the maintenance dose had been reached. One test pen was to be supplied per subject at the screening visit in order to ensure the subject's willingness and ability to self-inject. The test pen contained semaglutide placebo, solution for injection, 1.5 mL prefilled PDS290 pen-injector and was to be administered once. The PDS290 pen-injector for semaglutide is a prefilled pen integrated with a 1.5 mL cartridge containing semaglutide 1.34 mg/mL and is designed to be used with NovoFine®, NovoFine® Plus and NovoTwist® disposable needles. Once weekly (same day of the week) administered by s.c. injection in thigh, abdomen or upper arm, at any time of the day.
- Semaglutide 1.0 mg/Week: Subjects randomised to semaglutide followed a fixed dose-escalation regimen. The maintenance dose of 1.0 mg was to be reached after 4 doses (4 weeks) of 0.25 mg, followed by 4 doses (4 weeks) of 0.5 mg semaglutide. Doses could not be changed during the trial after the maintenance dose had been reached. One test pen was to be supplied per subject at the screening visit in order to ensure the subject's willingness and ability to self-inject. The test pen contained semaglutide placebo, solution for injection, 1.5 mL prefilled PDS290 pen-injector and was to be administered once. The PDS290 pen-injector for semaglutide is a prefilled pen integrated with a 1.5 mL cartridge containing semaglutide 1.34 mg/mL and is designed to be used with NovoFine®, NovoFine® Plus and NovoTwist® disposable needles. Once weekly (same day of the week) administered by s.c. injection in thigh, abdomen or upper arm, at any time of the day.
- Insulin Glargine: Subjects on insulin glargine were to start on 10 IU s.c. injected OD. The insulin dose adjustment had to aim to reach a pre-breakfast FPG of 4.0 to <5.5 mmol/L (71- <100 mg/dL). Once daily solution for injection in a 3 mL pre-filled SoloStar® pen to be administered in the thigh, abdomen or upper arm, at any time of the day
Period: Overall Study
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Started | 362 | 360 | 360
Completed | 335 | 341 | 342
Not Completed | 27 | 19 | 18
Not completed — Withdrawal by Subject | 11 | 7 | 8
Not completed — Death | 2 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — No reason for withdrawal | 12 | 11 | 7

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects who had received at least one dose of randomised semaglutide (s.c.) or insulin glargine. Subjects in the FAS contributed to the evaluation based on the treatment assigned at randomisation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine | Total
Number analyzed (Participants) | 362 | 360 | 360 | 1082
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.3) | 56.7 (10.4) | 56.2 (10.6) | 56.5 (10.4)
Age, Customized [Number; unit: Participants]
  18-64 years | 278 | 281 | 281 | 840
  65-74 years | 72 | 61 | 67 | 200
  75-84 years | 12 | 18 | 12 | 42
  >=85 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 178 | 165 | 508
  Male | 197 | 182 | 195 | 574
HbA1c [Mean (Standard Deviation); unit: percentage] | 8.13 (0.85) | 8.25 (0.94) | 8.13 (0.88) | 8.17 (0.89)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 172.4 (50.52) | 179.2 (53.74) | 174.2 (49.06) | 175.3 (51.18)
Body weight [Mean (Standard Deviation); unit: kg] | 93.73 (21.39) | 94.00 (22.48) | 92.61 (21.52) | 93.45 (21.79)
Diastolic Blood pressure [Mean (Standard Deviation); unit: mmHg] | 79.67 (8.04) | 80.32 (8.32) | 79.78 (9.20) | 79.72 (8.53)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131.57 (14.06) | 132.21 (16.05) | 132.38 (15.77) | 132.06 (15.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline
Description: Change in HbA1c from baseline to week 30.
Time Frame: Week 0, week 30
Population: The full analysis set (FAS) included all randomised subjects who had received at least one dose of randomized semaglutide (s.c.) or insulin glargine. Subjects in the FAS contributed to the evaluation based on the treatment assigned at randomisation.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
percentage | -1.21 (0.05) | -1.64 (0.05) | -0.83 (0.05)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg/Week vs Insulin Glargine; The post baseline responses were analysed using a mixed model for repeated measurements with treatment , country and stratum as fixed factors and baseline value as covariate, all nested within visit; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the upper limit of the two-sided 95% confidence interval for the estimated treatment difference between semaglutide 1.0 mg and insulin glargine was below the pre-specified non-inferiority margin (0.3 %); p < 0.0001, Mixed Models Analysis; Treatment difference = -0.81, 95% CI 2-sided [-0.96 to -0.67]
Statistical Analysis 2: Comparison: Semaglutide 0.5mg/Week vs Insulin Glargine; The post baseline responses were analysed using a mixed model for repeated meausrements with treatment, country and stratum value as covariate, all nested within visit; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the upper limit of the two-sided 95 % confidence interval for the estimated treatment difference between semaglutide 0.5 mg and insulin glargine was below the pre-specified non-inferiority margin (0.3%); p < 0.0001, Mixed Models Analysis; Treatment difference = -0.38, 95% CI 2-sided [-0.52 to -0.24]

2. Secondary Outcome: Change in Body Weight From Baseline
Description: Change in body weight from baseline to week 30.
Time Frame: Week 0, week 30
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
Kg | -3.47 (0.24) | -5.17 (0.24) | 1.15 (0.23)

3. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline
Description: Change in fasting plasma glucose from baseline to week 30.
Time Frame: Week 0, week 30
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
mg/dL | -36.74 (2.14) | -49.21 (2.15) | -38.18 (2.03)

4. Secondary Outcome: Change in Diastolic Blood Pressure.
Description: Change in diastolic blood pressure from baseline to week 30.
Time Frame: Week 0, week 30
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
mmHg | -1.38 (0.43) | -0.98 (0.44) | -1.44 (0.41)

5. Secondary Outcome: Change in Systolic Blood Pressure.
Description: Change in systolic blood pressure from baseline to week 30.
Time Frame: Week 0, week 30
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
mmHg | -4.65 (0.72) | -5.17 (0.73) | -1.68 (0.68)

6. Secondary Outcome: Change in Patient Reported Outcome (PRO) Questionnaire, Questionnaire SF-36v2™
Description: The Short Form (SF)-36v2™ patient reported outcomes (PRO) questionnaire was used to assess the subject's overall health related quality of life (HRQoL. PRO questionnaire (SF-36v2™) measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to a norm-based score using a T-score transformation in order to obtain a direct interpretation in relation to the distribution of the scores in the 1998 U.S. general population. The (SF-36v2™) values displayed are the estimated mean change from baseline to week 30.
Time Frame: Week 0, week 30
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
T-scores
  Bodily pain | 0.95 (0.51) | 1.76 (0.51) | 0.90 (0.48)
  General Health | 1.95 (0.38) | 2.78 (0.38) | 1.63 (0.36)
  Mental Component summary, MCS | 1.23 (0.47) | 1.33 (0.47) | 0.25 (0.44)
  Mental Health | 1.69 (0.46) | 1.17 (0.47) | 0.54 (0.44)
  Physical Component summary, PCS | 1.18 (0.36) | 2.09 (0.36) | 1.18 (0.34)
  Physical Functioning | 1.64 (0.43) | 1.49 (0.43) | 0.69 (0.41)
  Role-emotional | 0.88 (0.54) | 1.73 (0.54) | 0.06 (0.51)
  Role-physical | 0.90 (0.46) | 1.97 (0.46) | 0.78 (0.43)
  Social functioning | 1.13 (0.48) | 1.04 (0.48) | 0.36 (0.45)
  Vitality | 1.71 (0.46) | 2.09 (0.46) | 0.95 (0.44)

7. Secondary Outcome: Change in Patient Reported Outcome Questionnaires. (PROs), Diabetes Treatment Satisfaction Questionnaire (DTSQs)
Description: The Diabetes Treatment Satisfaction Questionnaire (DTSQs) questionnaire was to be used to assess a subject's treatment satisfaction. This questionnaire contained 8 components and measured the treatment for diabetes (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings regarding treatment. The value presented is the 'Treatment Satisfaction' summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction. The values displayed are the estimated mean change from baseline to week 30.
Time Frame: Week 0, week 30
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
Score on a scale | 4.86 (0.28) | 5.37 (0.29) | 3.99 (0.27)

8. Secondary Outcome: Subjects Who Achieve HbA1c ≤6.5% (48 mmol/Mol), American Association of Clinical Endocrinologists (AACE)
Description: Subjects who achieve HbA1c ≤6.5% (48 mmol/mol), American Association of Clinical Endocrinologists (AACE) after 30 weeks of treatment
Time Frame: After 30 weeks treatment
Population: as for baseline characteristics
Measure: Number; unit: Count of participants
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Number analyzed (Participants) | 362 | 360 | 360
Count of participants
  Yes | 135 | 195 | 63
  No | 227 | 165 | 297

ADVERSE EVENTS:
Time Frame: All adverse events presented here are treatment emergent adverse events (TEAE). A TEAE included events that had onset date (or increase in severity) on or after the first day of exposure (week 0) to randomised treatment (week 0-30 treatment period) and no later than the follow-up visit during the on-treatment observation period (date of last dose + 42 days).
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that had onset date (or increased in severity) during the 'on-treatment' observation period.
Arm/Group | Semaglutide 0.5mg/Week | Semaglutide 1.0 mg/Week | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 22/362 | 17/360 | 18/360
Other Adverse Events (participants affected / at risk) | 172/362 | 192/360 | 107/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5mg/Week (N=362) | Semaglutide 1.0 mg/Week (N=360) | Insulin Glargine (N=360)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal graft rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumocephalus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5mg/Week (N=362) | Semaglutide 1.0 mg/Week (N=360) | Insulin Glargine (N=360)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 18 (20) | 7 (10)
Decreased appetite (Metabolism and nutrition disorders) | 25 (34) | 23 (23) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 59 (67) | 69 (118) | 16 (18)
Dyspepsia (Gastrointestinal disorders) | 12 (24) | 24 (39) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 19 (20) | 3 (4)
Headache (Nervous system disorders) | 19 (40) | 23 (33) | 20 (26)
Lipase increased (Investigations) | 36 (39) | 30 (32) | 15 (17)
Nasopharyngitis (Infections and infestations) | 45 (58) | 29 (37) | 44 (51)
Nausea (Gastrointestinal disorders) | 77 (101) | 80 (117) | 12 (15)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 14 (16) | 24 (25)
Vomiting (Gastrointestinal disorders) | 24 (28) | 37 (119) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator (s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for upto 60 days to protect intellectual property.